CLINICAL TRIAL: NCT07398859
Title: A Multi-center, Open-label, Phase II, Single-arm Clinical Study Evaluating the Safety and Efficacy of TQH2722 Injection Combined With Background Treatment in Subjects With Seasonal Allergic Rhinitis
Brief Title: Clinical Study on TQH2722 Injection Combined With Background Therapy for Seasonal Allergic Rhinitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQH2722-II-06
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQH2722 injection (Experimental): Injection combined with TQH2722, 2 weeks as a treatment cycle.
  Interventions: Drug: TQH2722 injection

INTERVENTIONS:
Drug: TQH2722 injection — TQH2722 injection is a humanized monoclonal antibody targeting interleukin-4 receptor alpha (IL-4Rα).

SUMMARY:
This study is a multicenter, open-label, Phase II, single-arm clinical trial, with a planned enrollment of 200 to 300 subjects. Its primary objective is to evaluate the safety and efficacy of TQH2722 injection in the treatment of seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75, with no gender restrictions.
* Diagnosed with seasonal allergic rhinitis.
* Positive allergen test result.
* The subjects have sufficient exposure to pollen during the pollen season.
* The subject's medical history indicates that the subject had poor control of Seasonal Allergic Rhinitis (SAR) symptoms during the previous pollen season or the subject was dissatisfied with the subjective symptom control.
* Screen for subjects who have a morning iTNSS score of ≥4 on the day of screening; at baseline visit, have a morning iTNSS score of ≥4, and have an average rTNSS score of ≥4 over the past 6 days.
* Good compliance during screening/induction period.
* Subjects with comorbid asthma should have stable medication use before the screening period and have their asthma condition assessed as stable by the investigator or specialist.
* The subjects voluntarily joined this study, signed the informed consent form, and exhibited good compliance.
* The subjects and their partners agree to take effective contraceptive measures throughout the entire study period (from the signing of the Informed Consent Form (ICF) to 3 months after the last administration of the trial drug).

Exclusion Criteria:

* Any abnormal laboratory test value during the screening period or randomization.
* Any disease that researchers consider to be unstable and may affect the patient's safety throughout the entire study period, or affect the study results or their interpretation, or hinder the patient's ability to complete the entire study process.
* Patients with active autoimmune diseases.
* Known or suspected immunosuppressants.
* Subjects with active malignant tumors or a history of malignant tumors.
* Screen for individuals with a history of active tuberculosis within the previous 12 months.
* During the screening period, there is active hepatitis, or the presence of human immunodeficiency virus antibody (Anti-HIV) positivity, or syphilis treponema antibody (Anti-TP) positivity.
* Screen for cases diagnosed with helminthic parasitic infections within the previous 6 months, who have not undergone standard treatment or have experienced ineffective standard treatment.
* Subjects who have received specific medications or undergone any nasal or sinus surgery within the specified timeframe.
* Intravenous immunoglobulin (IVIG) therapy and/or plasma exchange within 30 days before screening.
* Screen subjects who have used monoamine oxidase inhibitors within the previous 14 days.
* Initiate allergen immunotherapy within 3 months prior to screening.
* Screen for individuals who have received attenuated live vaccines within the previous 4 weeks or plan to receive attenuated live vaccines during the study period.
* Screen for systemic Chinese herbal preparations used for the treatment of AR with short- or medium-acting systemic glucocorticoids within 4 weeks, or screen for long-acting Systemic Corticosteroids (SCS) received within the previous 6 weeks.
* Suffering from chronic active or acute infection within 2 weeks before screening or during the screening and import period.
* Patients with concomitant asthma should be excluded if they meet any of the following conditions: a. forced expiratory volume in one second (FEV1) ≤ 50% of the predicted normal value; b. acute exacerbation of asthma within 90 days prior to screening; c. currently using fluticasone propionate at a daily dose of >1000 μg/day or equivalent doses of other inhaled corticosteroids; d. assessed by the investigator or specialist as having unstable asthma.
* The subject has a concomitant disease that renders them unable to complete the screening period assessment or evaluate the primary efficacy endpoint.
* Suffering from malignant and benign tumors in the nasal cavity.
* Subjects with perennial allergic rhinitis (PAR) who are allergic to pet hair.
* Unable to use nasal corticosteroid sprays or antihistamines.
* Have a history of systemic allergy to any biological agents.
* Women who are pregnant or breastfeeding.
* Individuals who abuse alcohol, use drugs, and have known drug dependency.
* History of major organ transplantation or hematopoietic stem cell/bone marrow transplantation.
* According to the researcher's judgment, there are any medical or psychiatric symptoms that may put the subjects at risk, interfere with their participation in the study, or interfere with the interpretation of the study results.
* The forced expiratory volume in one second (FEV1) of the subject is less than or equal to 50% of the predicted normal value.
* Other reasons why the researcher believes it is inappropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with incidence of adverse event | Baseline up to 4 weeks
  Adverse events occurring during treatment.

SECONDARY OUTCOMES:
Number of subjects with incidence of serious adverse event | Baseline up to 4 weeks
  Serious adverse event occurring during treatment.
Number of subjects with incidence of abnormality check indicators | Baseline up to 4 weeks
  Number of subjects with incidence of abnormality check indicators: Abnormal examination indicators occurred during treatment.
Retrospective nasal symptom score after treatment for 2 weeks | Baseline up to 2 weeks
  The average change in the retrospective total nasal symptom score (rTNSS) per day over 2 weeks of treatment compared to baseline. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Retrospective nasal symptom score after treatment for 4 weeks | Baseline up to 4 weeks
  The average change in the retrospective total nasal symptom score (rTNSS) per day over 4 weeks of treatment compared to baseline. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Mean daily morning retrospective total nasal symptom score | Baseline up to 2 and 4 weeks
  Mean change from baseline in the morning retrospective total nasal symptom score (AM rTNSS) at 2 weeks and 4 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Mean daily retrospective total nasal symptom score at night | Baseline up to 2 and 4 weeks
  Mean change from baseline in the Post-Medication Reviewed Total Nasal Symptom Score (PMrTNSS) at night per day at 2 weeks and 4 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Total instantaneous nasal symptom score before medication in the morning every day | Baseline up to 2 and 4 weeks
  Mean change from baseline in instantaneous total nasal symptom score (iTNSS) before medication administration in the morning, for each day during the 2-week and 4-week treatment periods. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Daily retrospective total nasal symptom score | Baseline up to 2 and 4 weeks
  Mean percentage change from baseline in daily rTNSS at 2 weeks and 4 weeks of treatment.
Total instantaneous nasal symptom score before medication in the morning every day | Baseline up to 2 and 4 weeks
  Mean percentage change from baseline in iTNSS before medication administration in the morning, for each day during the 2-week and 4-week treatment periods.
Daily retrospective scoring of individual nasal symptoms | Baseline up to 2 and 4 weeks
  Mean change from baseline in daily retrospective nasal single symptom scores at 2 weeks and 4 weeks of treatment.
Daily retrospective nasal single symptom score during daytime | Baseline up to 2 and 4 weeks
  Mean change from baseline in retrospective daytime (AM) nasal individual symptom scores (rhinorrhea, nasal congestion, nasal itch, and sneezing) at 2 weeks and 4 weeks of treatment.
Daily retrospective nasal single symptom score during night | Baseline up to 2 and 4 weeks
  Mean change from baseline in retrospective nasal individual symptom (rhinorrhea, nasal congestion, nasal itch, and sneezing) scores at night (PM) at 2 weeks and 4 weeks of treatment.
Daily retrospective total score of ocular symptoms | Baseline up to 2 and 4 weeks
  Mean change from baseline in the retrospective Total Ocular Symptom Score (rTOSS) at 2 weeks or 4 weeks of treatment.
Total score of retrospective ocular symptoms during daytime each day | Baseline up to 2 and 4 weeks
  Mean change from baseline in the total daytime retrospective ocular symptom score (AM rTOSS) at 2 weeks and 4 weeks of treatment.
Total score of retrospective ocular symptoms each night | Baseline up to 2 and 4 weeks
  The average change in the retrospective total ocular symptom score (PM rTOSS) at night compared to baseline after 2 weeks and 4 weeks of treatment.
Total score of instantaneous ocular symptoms before medication in the morning every day | Baseline up to 2 and 4 weeks
  Mean change from baseline in instantaneous total ocular symptom score (iTOSS) before medication administration in the morning, at 2 weeks and 4 weeks of treatment.
Daily retrospective total score of ocular symptoms | Baseline up to 2 and 4 weeks
  Mean percentage change in total retrospective ocular symptom score from baseline at 2 weeks and 4 weeks of treatment, respectively.
Total score of instantaneous ocular symptoms before medication each morning | Baseline up to 2 and 4 weeks
  Mean percentage change from baseline in total ocular symptom score immediately before medication administration in the morning, for the 2-week and 4-week treatment periods.
Daily retrospective scoring of individual ocular symptoms | Baseline up to 2 and 4 weeks
  Mean change in individual ocular symptom scores from baseline to 2 weeks and 4 weeks after treatment, retrospectively assessed daily.
Daily retrospective scoring of individual ocular symptoms during the day | Baseline up to 2 and 4 weeks
  Mean change from baseline in retrospective ocular symptom scores during daytime (AM) on each day at 2 weeks and 4 weeks of treatment.
Nightly retrospective scoring of individual ocular symptoms | Baseline up to 2 and 4 weeks
  Mean change from baseline in retrospective ocular symptom scores at night (PM) at 2 weeks and 4 weeks of treatment
Quality of Life Questionnaire Score for Patients with Allergic Rhinitis | Baseline up to 2 and 4 weeks
  The change in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scores from baseline for patients with allergic rhinitis after 2 weeks and 4 weeks of treatment.
Daily retrospective total score of nasal symptoms | Baseline up to 2 and 4 weeks
  The area under the curve representing the average change in the retrospective total nasal symptom score (rTNSS) from baseline, calculated for each day during the 2-week and 4-week treatment periods.
Blood eosinophil count and percentage | Baseline up 12 weeks
  Changes in eosinophil count and percentage from baseline, as well as the percentage of change, at each evaluation visit point.
Serum total immunoglobulin E concentration | Baseline up 12 weeks
  The changes in serum total immunoglobulin E concentration and the percentage of change from baseline at each evaluation visit point.
Forced expiratory volume in 1 second (FEV1) before bronchodilator administration (BD) in subjects with concomitant asthma | Baseline up 12 week
  The change in forced expiratory volume in one second (FEV1) relative to baseline before the use of bronchodilator (BD) in subjects with asthma across all visit points.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Hebei University Affiliated Hospital, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei PetroChina Central Hospital, Langfang, Hebei
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of science and technology, Wuhan, Hubei
  - Tongji Hospital of Tongji medical college of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Yan'an University Xianyang Hospital, Xi'an, Shaanxi
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Second People's Hospital of Chengdu, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Provincial Hospital of Chinese Medicine, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang